CLINICAL TRIAL: NCT02772042
Title: Effectiveness of Traction Manipulation of Upper Cervical Spine on Cervicogenic Dizziness
Brief Title: Traction Manipulation of Upper Cervical Spine on Cervicogenic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andoni Carrasco (Other)
Responsible Party: Sponsor-Investigator, Andoni Carrasco, PT, Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/0230
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Dizziness; Neck Pain
Keywords: Manual Therapy; Physiotherapy; Manipulation
MeSH Terms: conditions — Dizziness; Neck Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Investigators will performed traction manipulation of those articulations of upper cervical spine with indication for this treatment. Before manipulation soft tissue techniques will be applied in order to prepare the joint. After manipulation the patient rest in supine position. The intervention will have a duration of 10 minutes.
  Interventions: Other: Intervention Group
- Control Group (Other): The patient of the control group maintain the supine position for 10 minutes.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group
  Arms: Intervention Group
Other: Control Group
  Arms: Control Group

SUMMARY:
Manual therapy reduces symptoms in patients with cervicogenic dizziness. The mobilization and manipulation of upper cervical spine are the most popular treatment in this patients. The International Federation of Orthopaedic Manipulative Physical Therapists suggest different recommendations for the safety application of manual therapy techniques in the upper cervical spine, traction manipulation techniques complies with this conditions. However, there isn´t investigation about the effect of traction manipulation in patients with cervicogenic dizziness. The aim of this study is to investigate the effects of traction manipulation in dizziness intensity, range of motion of cervical spine and quality of life on patients with cervicogenic dizziness.

ELIGIBILITY:
Inclusion Criteria:

* Dizziness associated with neck stiffness and/or neck pain.
* Hypomobility of upper cervical spine.
* Sing the informed consent form.

Exclusion Criteria:

* Contraindications for Traction manipulation.
* Pending litigation or legal claim.
* Poor language and communication skills making difficult to understand the informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change of baseline in Dizziness Intensity (100mm VAS) at 1 week and 1 month | Baseline- 1 week- 1 month

SECONDARY OUTCOMES:
Change of baseline in range of motion of cervical spine change (Tool: Cervical range of motion) | Baseline- 1 week- 1 month
Change of baseline in upper cervical spine range of motion (Tool: Cervical range of motion) | Baseline- 1 week- 1 month
Change of baseline in dizziness Handicap Inventory (questionnaire) | Baseline- 1 week- 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Andoni Carrasco, Pt, Principal Investigator — Unidad de Investigación en Fisioterapia. Universidad de Zaragoza
Locations (1):
- Unidad de Investgación en Fisioterapia. Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No